CLINICAL TRIAL: NCT02295891
Title: Microwave Energy-induced Thermolysis of Axillary Apocrine Glands and Hair Follicles Will Result in Improvement of Secondary Psychopathology Related to Hyperhidrosis.
Brief Title: Miradry Treatment for Focal Axillary Hyperhidrosis
Acronym: MiraDry Tx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was inactive and no continuing review was submitted, resulting in its expiration and termination
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00036743
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Axillary Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MiraDry ® treatment (Experimental): MiraDry ® is the trademarked name of a non-invasive thermolytic technology which utilizes a microwave energy-based mechanism targeted for eccrine gland reduction at the dermal-fat interface.
  Each participant will be scheduled two MiraDry ® treatment appointments approximately three months apart.
  Interventions: Device: MiraDry ®

INTERVENTIONS:
Device: MiraDry ® — Non-invasive thermolytic technology which utilizes a microwave energy-based mechanism targeted for eccrine gland reduction at the dermal-fat interface

SUMMARY:
Primary hyperhidrosis is a pathological condition characterized by the idiopathic and excessive secretion of sweat beyond normal physiological demand and is localized at particular foci such as the face, axilla, palms of the hands, and soles of the feet. Patients seeking medical attention for hyperhidrosis often report disruptions to their professional and/or social lives due to sweating and subsequently experience many psychosocial difficulties, such as anxiety, social phobia, and depression. Therefore, a psychiatric explanation of causality is frequently offered for these patients during diagnosis. Excessive sweating is often mistakenly interpreted as a symptom of an anxiety disorder and can be cause for social embarrassment, exacerbating emotional stress and social avoidance. As currently constituted, the treatment of secondary psychosocial symptoms in primary hyperhidrosis is poorly understood and requires further investigation.

DETAILED DESCRIPTION:
Primary Objective:

1. To evaluate the effectiveness of the miraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis.

   Secondary Objectives:
2. To characterize the outcomes of and clinical response to the MiraDry ® treatment system with respect to the aforementioned criteria.
3. To compare the results of non-invasive miraDry ® treatment system to the existing surgical correction with respect to the aforementioned criteria.

ELIGIBILITY:
Inclusion Criteria:

This study will recruit patients diagnosed with focal hyperhidrosis with a known diagnosis of primarily axillary localization.

We will only enroll patients available for both treatment visits. Availability for follow-up visit is optional.

Only patients between the ages of 18 and 29 years when the first HHIQ is administered will be eligible.

The upper age limit was so determined because patients over 29 years often present with psychopathology which is far more recalcitrant to correction of any kind regardless of effectiveness because of the duration of the condition.

The lower age limit was so determined because 18 years and up are the ages for which the miraDry ® procedure has been approved for use by the FDA.

All participants will be screened using the Hyperhidrosis Disease Severity Scale (HDSS).

Only patients reporting their condition as a 3 out of 4 or higher on the HDSS will be eligible for study because preliminary data suggests effective detection of psychological changes only at higher reported levels of sweating severity.

A patient's previous non-invasive treatment course, including but not limited to prescription of psychiatric medication and topical therapies, will not justify exclusion from this study.

Exclusion Criteria:

Patients who are unable to provide informed consent, have known allergies to lidocaine, hibiclens with 4% chlorhexidine, and/or epinephrine, are pregnant (as determined by self-reporting), are unable to take oral antibiotics or antiseptic washes, have heart pacemakers or other electronic device implants, and who need supplemental oxygen are not eligible to participate in this study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brock, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who have focal hyperhidrosis with a known diagnosis of primarily axillary localization were recruited from both the Johns Hopkins Department of Dermatology and Thoracic Surgery. The recruitment of these patients will occur during normal appointments and clinic visits at Johns Hopkins Hospital.
Pre-assignment Details: Total 31 patients signed consents-
  * 7 of the 31 consented but never scheduled 1st procedure and were not assigned to the arm
  * 24 patients were assigned to the arm
Groups:
- MiraDry ® Treatment Group: MiraDry ® is the trademarked name of a non-invasive thermolytic technology which utilizes a microwave energy-based mechanism targeted for eccrine gland reduction at the dermal-fat interface.
  Each participant will be scheduled two MiraDry ® treatment appointments approximately three months apart
Period: Overall Study
Arm/Group | MiraDry ® Treatment Group
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data collected for participants who had at least 1 psychological evaluation and 1 MiraDry treatment appointment
Arm/Group | MiraDry ® Treatment Group
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants]
  18 to 29 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
hyperhidrosis in primarily axillary localization [Count of Participants; unit: Participants] | 24

OUTCOME MEASURES:

1. Primary Outcome: Disease Severity as Assessed by the Hyperhidrosis Disease Severity Scale (HDSS)
Description: To evaluate the effectiveness of the miraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis. Patients will be asked to complete the Hyperhidrosis Disease Severity Scale (HDSS). HDSS assigns a point value where severity is scored: Minimal (1)=My sweating is never noticeable and never interferes with my daily activities to most severe score is: (4)=My sweating is intolerable and always interferes with my daily activities. Lower point values are considered better and higher point values are considered worse.
Time Frame: Baseline, 6 months, 1 Year
Population: Participants with data collected are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MiraDry ® Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 3.46 (0.51)
  6 months: number analyzed (Participants) | 22
  6 months | 2.5 (.96)
  1 year: number analyzed (Participants) | 20
  1 year | 2.05 (.83)

2. Primary Outcome: Quality of Life as Assessed by the Dermatology Quality of Life Index
Description: To evaluate the effectiveness of the miraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis. Patients will be asked to complete the Dermatology Quality of Life Index. Total score range from 0-30, a higher score indicating more impairment on the participant's quality of life
Time Frame: Baseline, 6 months, 1 Year
Population: Participants with data collected are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MiraDry ® Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 12.92 (5.47)
  6 months: number analyzed (Participants) | 22
  6 months | 6.25 (5.74)
  1 year: number analyzed (Participants) | 20
  1 year | 3.68 (4.31)

3. Primary Outcome: Social Phobia as Assessed by the Social Phobia Inventory (SPIN)
Description: To evaluate the effectiveness of the miraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis. Patients will be asked to complete the Social Phobia Inventory (SPIN) consisting of 17 questions to assess social phobia. The lowest possible score is 0 and the highest is 68. A score of 19 or more on the SPIN suggests social phobia or social anxiety disorder. A lower score, or reduction in score, is better.
Time Frame: Baseline, 6 months, 1 Year
Population: Participants with data collected are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MiraDry ® Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 28.83 (12.04)
  6 months: number analyzed (Participants) | 22
  6 months | 17.91 (14.34)
  1 year: number analyzed (Participants) | 20
  1 year | 15.90 (11.87)

4. Primary Outcome: Anxiety as Assessed by the Zung Self-rating Anxiety Scale (ASL)
Description: To evaluate the effectiveness of the miraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis. Patients will be asked to complete the Zung Self-rating Anxiety Scale (ASL). The score range is 20-80: 20-44 Normal Range, 45-59 Mild to Moderate Anxiety Levels, 60-74 Marked to Severe Anxiety Levels, 75-80 Extreme Anxiety Levels.
Time Frame: Baseline, 6 months, 1 Year
Population: Participants with data collected are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MiraDry ® Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 45.67 (10.22)
  6 months: number analyzed (Participants) | 22
  6 months | 30.96 (7.64)
  1 year: number analyzed (Participants) | 20
  1 year | 27.50 (11.87)

5. Primary Outcome: Functioning as Assessed by the Achenbach Self Report (ASR)
Description: To evaluate the effectiveness of the MiraDry ® treatment system for psychosocial functioning in patients heavily affected by axillary hyperhidrosis. Patients will be asked to complete the Achenbach Self Report, with a score range of 0 to 240, with score of 65 being marked as concerning. A lower score correlates to better functioning.
Time Frame: Baseline, 6 months, 1 Year
Population: Participants with data collected are reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MiraDry ® Treatment
Number analyzed (Participants) | 24
score on a scale
  Baseline | 61.38 (12.68)
  6 months: number analyzed (Participants) | 22
  6 months | 53.75 (5.34)
  1 year: number analyzed (Participants) | 20
  1 year | 53.35 (4.29)

ADVERSE EVENTS:
Time Frame: Up to 24 months.
Groups:
- MiraDry ® Treatment Group: Patients who suffer from psychosocial symptoms related to axillary hyperhidrosis. Each patient is required to undergo 2 MiraDry treatments, 3 months apart. The patients are also required to complete 4 surveys at the initial appointment, and the same 4 again at follow up.
Arm/Group | MiraDry ® Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
Some patients had issues with the cost of the third round of treatments, if necessary. Sometimes the study team needed to reach out a few times in order to get all questionnaires completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT02295891/Prot_SAP_000.pdf
  • Informed Consent Form (2014-10-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02295891/ICF_001.pdf